CLINICAL TRIAL: NCT06580743
Title: Efficacy Verification in Early Diagnosis and Management of Lymphedema Through Home Body Water Analyzer
Status: Completed | Type: Observational
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Other Study IDs: PT-2024-32330
Record Dates: First submitted 2024-08-16; First posted 2024-08-30 (Actual); Last update posted 2025-10-01 (Actual); Status verified 2025-09

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Study group: breast cancer patients 1-12 months post surgery
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — This is an observational study

SUMMARY:
Breast cancer is the second most common cancer in women. One in five women who have been treated for breast cancer develop lymphedema. Lymphedema is a very common result of breast cancer and its treatment. Lymphedema is the build-up of fluid in tissues, which results in tissue swelling. The lymph system is a network of lymph vessels, tissues, and organs that carry extra fluid from your cells/tissues throughout the body. If this lymph fluid is not able to flow in the body how it should, there will be swelling which can lead to lymphedema. It can be classified into stages 0 to 3 depending on the severity of the condition. Stages 0 and 1 are reversible, and through early diagnosis and treatment, the recovery to the normal volume and normal skin status of arms can be possible. On the other hand, stage 2 or higher is irreversible, and tissue fibrosis progresses and cannot return to normal skin; therefore, it is important to detect early and start treatment.

This is an observational longitudinal study. Potential participants will be recruited for follow-up after breast cancer surgery. Only patients who fit the inclusion criteria will be considered for participation in the study and contacted by the healthcare provider. Standard of care will be used to guide any treatment needed by participants while they are part of the study.

ELIGIBILITY:
Inclusion Criteria:

* Adults 18 and over who are diagnosed with unilateral breast cancer.
* Unilateral lumpectomy, unilateral mastectomy, or simultaneous contralateral prophylatic mastectomy within 12 months of enrollment
* Axillary lymph node dissection or sentinel node biopsy within 12 months of enrollment
* Adjuvant or neoadjuvant chemotherapy and/or radiation therapy are allowed
* Breast cancer reconstruction completed or planned is allowed
* Study participants must own or have access to a smartphone, iPhone (IOS version 9.0 or above) or Android phone (Android 8.1 or above).

Exclusion Criteria:

* Bilateral breast cancer
* Previous history of breast cancer prior to current diagnosis.
* Existing diagnosis of lymphedema at the time of enrollment
* Cellulitis or other active infection at the time of enrollment
* Adults who are unable to consent.
* Pregnant women
* Prisoners
* Individuals under the age of 18 years old
* Individuals who are illiterate
* Individuals who lack the capacity to consent
* Non-English speakers
* Individuals with medical implant devices such as pacemakers, or essential support devices such as patient monitoring systems.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: check inclusion criteria
Sampling Method: Non-Probability Sample
Enrollment: 52 (Actual)
Dates: Start 2024-06-12 (Actual); Primary Completion 2025-09-30 (Actual); Study Completion 2025-09-30 (Actual)

PRIMARY OUTCOMES:
Measurement of impedances and extracellular water (ECW) ratio | 3, 6, 9, and 12 months
  Measurement of impedances and extracellular water (ECW) ratio between affected and unaffected sides at initial visit using the clinical and home units (InBody 770 and InBody BWA ON).
  Inbody BWA 770 Timeline: baseline, 3, 6, 9, 12 month Inbody BWA ON Timeline: 2x/day x 12 months

SECONDARY OUTCOMES:
Measurement of impedances and extracellular water (ECW) ratio | 3, 6, 9, and 12 months
  Measurement of impedances and extracellular water (ECW) ratio between affected and unaffected sides at 3, 6, 9, and 12 months using the clinical and home units.
attitudes | 12 months
  Measure qualitative responses through exit interviews with participants to learn their attitudes toward their evaluation with the home BIA home device at 12 months.
Bilateral upper extremity shoulder goniometric range of motion measurements | baseline, 3, 6, 9, and 12 months
  measured in degrees
Bilateral upper extremity girth circumference measurements | baseline, 3, 6, 9, and 12 months
  measured in centimeters
Impact of lymphedema | baseline, 3, 6, 9, and 12 months
  Lymphedema Life Impact Scale questionnaire LLIS consists of 18 questions divided into physical, functional, and psychosocial domains. The questions are rated from 0-4 with 0 being no symptoms and 4 being severe symptoms.
Disabilities | baseline, 3, 6, 9, and 12 months
  Disabilities of the Arm, Shoulder and Hand questionnaire The DASH consists of 30 items of disability/symptom scale, each scored from 1 to 5. The final score is converted to a scale of 0 to 100 (higher scores represent higher disability).
Skin/tissue assessment | baseline, 3, 6, 9, and 12 months
  Skin/Tissue Assessment: Items assessed include Axillary Web Syndrome (present or absent), presence of visible/palpable lymphedema (location and severity-min/mod/severe), Stemmer's sign (positive or negative).

CONTACTS AND LOCATIONS:
Overall Officials: Linda A Koehler, PhD, Principal Investigator — University of Minnesota
Locations (1):
- University of Minnesota, Minneapolis, Minnesota, United States